CLINICAL TRIAL: NCT04148729
Title: Effect of USG Guided ESP Block in Spinal Surgery
Brief Title: USG Guided ESP Block in Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Anesthesiologist, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP block in Spinal Surgery
Record Dates: First submitted 2018-08-01; First posted 2019-11-01 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain
Keywords: erector spinae plane block; postoperative analgesia; spinal surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both participants and anaesthesia providers will not know contain of the syringe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bupivacaine+lidocaine (Active Comparator): 15 ml bupivacaine+ 5 ml lidocaine will use for USG guided ESP block under general anaesthesia with Sevuflurane and remifentanil. This block will perform at the T10 level bilaterally after induction of anaesthesia at the prone position. The patients will receive Morphine 0.1 microgram/kg intravenously and diclofenac sodium 75 mg intramuscularly at the last 30th minute of surgery. Postoperative pain assessment will perform with VAS score. The rescue analgesic 0.4 mg/kg meperidine will be apply intravenously whenever the patient requested to the analgesic.
  Interventions: Drug: ESP block
- saline (Sham Comparator): In this group, the same volume saline will apply to the block region. The patients will receive Morphine 0.1 microgram/kg intravenously and diclofenac sodium 75 mg intramuscularly at the last 30th minute of surgery. Postoperative pain assessment will perform with VAS score.
  The rescue analgesic 0.4 mg/kg meperidine will be apply intravenously whenever the patient requested to the analgesic.
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: ESP block — Ultrasound guided ESP block will perform with 15 ml bupivacaine+ 5 ml lidocaine at the T10 level bilaterally. 0.1 microgram morphine (IV) and diclofenac sodium 75 mg intramuscularly will perform for postoperative analgesia.
  Arms: bupivacaine+lidocaine
Drug: Control Group — In this group Ultrasound guided ESP block will not perform. Postoperative analgesia will provide with 0.1 microgram morphine (IV) and diclofenac sodium 75 mg intramuscularly.
  Arms: saline

SUMMARY:
American Society of Anaesthesiologist physical status I-II, aged between 18-65, 40 patients which underwent lumbar spinal surgery will recruited to this study. These subjects will Ultrasound (USG) guided erector spinae block will perform at T10 level (bilaterally) to the all patient under general anaesthesia. 15 ml bupivacaine %0.5 and 5 ml lidocaine %2 will use for USG guided ESP block. 0.1 microgram/kg morphine will apply intravenously and diclofenac Na 75 mg intramuscularly will apply at last 30 minutes of surgery postoperative analgesia to all patients. Postoperative pain assessment will perform with visual analog scale (VAS)

DETAILED DESCRIPTION:
American Society of Anaesthesiologist physical status I-II, aged between 18-65, 40 patients which underwent lumbar spinal surgery will recruited to this study. The patients were randomly allocated into two groups (1:1), via a computer-generated randomization list. Ultrasound (USG) guided erector spinae block will perform at T10 level (bilaterally) to the 20 patients under general anaesthesia in Group E and same volume saline will apply to the ESP block region at T10 level for control group (Group C). Total intravenous anaesthesia (propofol+remifentanil) will perform to the all patients. 15 ml bupivacaine %0.5 and 5 ml lidocaine %2 will use for USG guided ESP block. 0.1 microgram/kg morphine intravenously and diclofenac Na 75 mg intramuscularly will apply for postoperative analgesia to the all patients at last 30 minutes of surgery. Postoperative pain assessment will perform with visual analog scale (VAS). VAS, morphine consumption and complications will record. The rescue analgesic 0.4 mg/kg mepheridine will administer intravenously whenever the patient requested to the analgesic. Diclofenac sodium 75 mg will repeat to the all patients at the 12th of postoperative period, intramuscularly.

ELIGIBILITY:
Inclusion Criteria:

* accepting to participate the study
* ASA I-II patients
* The patients underwent spinal surgery

Exclusion Criteria:

* Non Volunteers
* ASA III and over
* Renal and hepatic failure
* Emergency surgical procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
11-point numerical rating scale score (NRS score) | up the postoperative 24th hours.
  Postoperative pain assessment will perform with 11-point numerical rating scale score and numerical scale point which described by resident will record. Higher points show that severe pain. 0 point shows no pain.10 point shows unbearable pain.

SECONDARY OUTCOMES:
Postoperative analgesic requirement | up the postoperative 24th hours.
  When the higher points numerical scale point (4<) observed, additional analgesics will apply. An than, totally consumption of rescue analgesic requirement (meperidine consumotion) will calculate.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova University, Adana, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No